CLINICAL TRIAL: NCT07346105
Title: An Expanded Access Program for Orca-T Products That Are Out of Specification for Commercial Release
Brief Title: Orca-T Expanded Access Program Study for Patients With Advanced Hematologic Malignancies
Status: Temporarily not available | Type: Expanded Access
Sponsor: Orca Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Orca-T OOS EAP
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancies; Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Myelodysplastic Syndrome; Mixed Phenotype Acute Leukemia
Keywords: Hematopoietic stem cell transplantation; Acute leukemia; Myelodysplastic syndromes; Matched related donor; Matched unrelated donor; Myelodysplastic syndrome
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Biphenotypic, Acute

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Orca-T — Orca-T that does not meet commercial release specifications

SUMMARY:
This study is not designed to test a hypothesis; rather, this study will provide patients with access to Orca-T if the commercial Orca-T product produced for them is deemed out of specification (OOS). Serious adverse events (SAEs) occurring during the safety reporting period (defined as the day the recipient receives the Orca-T HSPC drug product through day +365 after transplantation or until initiation of new anticancer therapy, whichever occurs sooner) will be reported.

ELIGIBILITY:
Inclusion Criteria:

Recipients in this EAP must meet all of the following criteria:

1. Commercial Orca-T was prescribed to the patient by their treating physician.
2. The final manufactured Orca-T does not meet the commercial release specifications or is delivered past expiry.
3. The final manufactured Orca-T is acceptable per joint assessment by Orca Bio and the treating physician, taking into account Orca Bio's release criteria.
4. Remanufacturing (ie, repeat leukapheresis and manufacturing) is not clinically appropriate per the treating physician's assessment.
5. Recipient must be deemed medically fit and stable to receive Orca-T infusions per the treating physician's evaluation.

Exclusion Criteria:

Recipients with any medical condition identified by the treating physician that may impact the safety or outcomes of the recipient in relation to treatment with Orca-T will not be eligible.

Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Background] Meyer E, Salhotra A, Gandhi A, Pantin J, Patel SS, Hoeg RT, Gomez-Arteaga A, Faramand RG, Tamari R, Waller EK, Kosuri S, Jimenez Jimenez AM, Holter-Chakrabarty J, Dholaria B, Chen YB, Hamilton BK, Magenau JM, Eghtedar A, Murray JM, Pavlova A, Fernhoff NB, McClellan JS, Killian S, Li A, Negrin RS, Oliai C. Orca-T versus allogeneic hematopoietic stem cell transplantation (PRECISION-T): a multicenter, randomized phase 3 trial. Blood. 2025 Dec 12:blood.2025031313. doi: 10.1182/blood.2025031313. Online ahead of print. PMID 41385341